CLINICAL TRIAL: NCT07205250
Title: WesternTheaterCommand
Brief Title: Aspirin for Prevention of Stroke After Endovascular Aortic Arch Repair: a Multicenter, Double-Blind, Randomized Controlled Trial
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The General Hospital of Western Theater Command (Other)
Responsible Party: Principal Investigator, siyi He, Deputy Chief Physician, Associate Professor, The General Hospital of Western Theater Command
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: hesiyi WesternTheaterCommand
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Type B or Non-A Non-B Aortic Dissection;Thoracic Aortic Aneurysm
Keywords: aspirin; stroke; endovascular aortic arch repair; prevention
MeSH Terms: conditions — Stroke | interventions — Tablets; Taste; Smell

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, double-blind, randomized, placebo-controlled, parallel-group clinical trial. Using a parallel-group design, participants are randomly assigned to one of three groups: three aspirin groups with different treatment durations (3 months, 6 months, 1 year). For the three-month and six-month aspirin groups, placebo administration will be maintained after completing the assigned treatment duration. All three groups proceed with the intervention concurrently. The study uses pre-defined efficacy endpoints to measure and evaluate outcomes synchronously.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study employs a double-blind method with a two-level blinding system. The core principle is the isolation of key roles and the withholding of information.
  Blinding Personnel / Drug Managers: The blinding personnel or drug managers are aware that Drug A is the investigational drug (aspirin) and Drug B is the placebo; however, they have no contact with study participants and do not participate in efficacy or safety assessments.
  Investigators / Assessors / Participants: Are responsible for the treatment, follow-up, and assessment of participants but are unaware of the specific identity of Drug A and Drug B (i.e., they do not know which is the investigational drug and which is the placebo).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aspirin 3-month group (Experimental): Patients in the Aspirin 3-month group will begin oral administration of enteric-coated aspirin tablets (100 mg once daily, Bayer Healthcare, specification: 100 mg/tablet) on the first postoperative day. The oral medication course will last for three months.Then receive placebo treatment for nine months.
  Interventions: Drug: enteric-coated aspirin tablets (100 mg once daily, Bayer Healthcare, specification: 100 mg/tablet); Other: a placebo with identical or similar appearance, taste, smell, and packaging to the aspirin tablets
- Aspirin 6-month group (Experimental): Patients in the Aspirin 6-month group will begin oral administration of enteric-coated aspirin tablets (100 mg once daily, Bayer Healthcare, specification: 100 mg/tablet) on the first postoperative day. The oral medication course will last for six months.Then receive placebo treatment for six months.
  Interventions: Drug: enteric-coated aspirin tablets (100 mg once daily, Bayer Healthcare, specification: 100 mg/tablet); Other: a placebo with identical or similar appearance, taste, smell, and packaging to the aspirin tablets
- Aspirin 1-year group (Experimental): Patients in the Aspirin 1-year group will begin oral administration of enteric-coated aspirin tablets (100 mg once daily, Bayer Healthcare, specification: 100 mg/tablet) on the first postoperative day. The oral medication course will last for one year.
  Interventions: Drug: enteric-coated aspirin tablets (100 mg once daily, Bayer Healthcare, specification: 100 mg/tablet)

INTERVENTIONS:
Drug: enteric-coated aspirin tablets (100 mg once daily, Bayer Healthcare, specification: 100 mg/tablet) — Patients are randomized into three groups using a random number table or lottery method: Aspirin 3-month group, Aspirin 6-month group, Aspirin 1-year group. Every group begin oral administration of aspirin enteric-coated tablets 100 mg once daily (qd) (Bayer Healthcare Co., Ltd., specification: 100 mg/tablet) on the first postoperative day. Aspirin 3-month group will receive the investigational drug for 3 months followed by placebo for 9 months; Aspirin 6-month group will receive the investigational drug for 6 months followed by placebo for 6 months; Aspirin 1-year will receive the investigational drug for 1 year).
Other: a placebo with identical or similar appearance, taste, smell, and packaging to the aspirin tablets — The placebo's smell, color, taste, and packaging are identical or very similar to the aspirin enteric-coated tablets (Shandong Xinhua Pharmaceutical Co., Ltd., one of the world's largest producers of aspirin API and finished dosage forms. The company has extensive tablet manufacturing experience and GMP certification. Specifications regarding the appearance [size, color, shape], weight, taste, etc., of the placebo have been clearly defined to ensure it is completely identical to the aspirin tablets used in the study).
  Arms: Aspirin 3-month group; Aspirin 6-month group

SUMMARY:
ABSTRACT Introduction Endovascular aortic arch repair (EAAR) and the endovascular reconstruction of arch branch vessels represent a new trend in managing aortic arch pathologies, due to advantages such as minimal invasiveness, rapid recovery, and fewer complications. However, stroke is a common and serious complication during EAAR procedures. Strategies for its prevention, including the question of whether antiplatelet therapy should be administered postoperatively, have not yet been reported.

Methods and analysis This project is designed as a prospective, multicenter, double-blind, randomized controlled trial. Patients undergoing Endovascular Aortic Arch Repair (EAAR) will be randomly assigned to three groups: aspirin treatment for 3 months, 6 months, or 1 year. All three groups will be followed up on for over one year. The primary endpoint is the incidence of postoperative stroke, while secondary endpoints include the patency rate of reconstructed supra-aortic branches, the incidence of major bleeding complications, EAAR-related complications, and the incidence of postoperative cognitive impairment. The study aims to evaluate the efficacy and safety of aspirin in preventing stroke after EAAR.

Furthermore, stratified analyses will be conducted based on factors such as reconstruction techniques, the number of reconstructed branch arteries, and the diameter of branch stents to explore their impact on stroke incidence post-EAAR. The clinical utility of aspirin in different subgroups will also be assessed to provide more precise and personalized treatment strategies for clinical practice.

Ethics and dissemination This study has been approved by the Western Theater Command General Hospital and will be conducted in accordance with the principles of the Declaration of Helsinki. Ethical approval has been obtained separately from all participating research centers.

STRENGTHS AND LIMITATIONS OF THIS STUDY Endovascular aortic arch repair (EAAR) and endovascular reconstruction of the aortic arch branches have emerged as a new trend in managing aortic arch pathologies, owing to advantages such as minimal invasiveness, rapid recovery, and fewer complications. Stroke is a common and serious complication during EAAR procedures; however, strategies for its prevention, including the need for postoperative antiplatelet therapy, have not been well documented.

This project aims to conduct a prospective, multicenter randomized controlled trial to evaluate the efficacy and safety of aspirin in preventing stroke following EAAR, thereby providing evidence for clinical decision-making and improving long-term patient outcomes. As the trial will be conducted in China, where the population is predominantly Han Chinese, the generalizability of the findings may be limited.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 years or older;
2. Diagnosed with type B or non-A non-B aortic dissection or thoracic aortic aneurysm according to the 2022 Chinese Expert Consensus on Stanford Type B Aortic Dissection;
3. Underwent total endovascular aortic arch repair at the participating center with concurrent intraoperative endovascular reconstruction of supra-arch branch arteries;
4. Signed the informed consent form and agreed to participate in this randomized controlled trial.

Exclusion Criteria

1. Patients with known allergies to aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs);
2. Patients with bleeding tendencies or active bleeding;
3. Patients who used medications affecting coagulation (e.g., warfarin, antiplatelet drugs) within 30 days before surgery;
4. Patients with a history of stroke;
5. Patients undergoing concurrent additional surgical procedures during the operation;
6. Patients with severe multi-organ dysfunction or other critical illnesses;
7. Patients unable to comply with study protocols or complete postoperative follow-up;
8. Patients participating in other drug or clinical studies that may interfere with the results of this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2028-01-20 (Estimated); Study Completion 2028-09-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative stroke. | After one year
  yes or no

SECONDARY OUTCOMES:
Patency rate of reconstructed branch vessels, | After one year
  yes or no
incidence of major postoperative bleeding complications, | After one year
  yes or no
incidence of complications related to endovascular aortic arch repair (e.g., thrombosis, bleeding, infection), | After one year
  yes or no
incidence of postoperative cognitive impairment. | After one year
  yes or no